CLINICAL TRIAL: NCT02182349
Title: Metabolism and Pharmacokinetics of a Single Dose of 240 mg [14C]-BI 201335 Given as Oral Solution to Healthy Male Volunteers at Steady State of BI 201335 NA Maintained With Oral Capsules of 240 mg BI 201335, a Phase I, Single-arm, Open-label Trial
Brief Title: Metabolism and Pharmacokinetics of Oral Solution of [14C]-BI 201335 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1220.33
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (1):
- BI 201335 NA (Experimental): multiple doses of BI 201335 NA soft gelatin capsule on days 1-8 and 11-15 and one single dose of [14C]-BI 201335 NA radiolabelled drug on day 9
  Interventions: Drug: BI 201335 NA soft gelatin capsule; Drug: [14C]-BI 201335 NA radiolabelled drug

INTERVENTIONS:
Drug: BI 201335 NA soft gelatin capsule
Drug: [14C]-BI 201335 NA radiolabelled drug

SUMMARY:
Study to determine the pharmacokinetics (PK) of BI 201335 and total radioactivity including excretion mass balance, excretion pathways and metabolism following the oral administration of [14C]-BI 201335 at steady state.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males according to a complete medical history, including a physical examination, vital signs (blood pressure, pulse rate), 12-lead ECG (electrocardiogram), and clinical laboratory tests
* Age 18 to 55 years, inclusive
* Body mass index 18.5 to 29.9 kg/m2, inclusive
* Nonsmoker
* Signed and dated written informed consent prior to admission to the study in accordance with GCP (Good Clinical Practice) and the local legislation

Exclusion Criteria:

* Any finding in the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, hormonal, psychiatric or neurological disorders (including all forms of epilepsy)
* Surgery of the gastrointestinal tract (except appendectomy)
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Subjects with Gilbert's Syndrome
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (>24 hours) within one month prior to administration of the trial drug
* Use of prescription medication, over-the-counter drugs or herbal preparations within 14 days prior to administration of the trial drug
* Participation in another trial with an investigational drug within two months prior to administration of the trial drug or during the trial
* History or evidence of habitual tobacco or nicotine use within six months prior to administration of the trial drug
* Alcohol abuse (more than 2 ounces of alcohol/day)
* Drug abuse in opinion of investigator
* Blood donation (more than 100 mL within four weeks prior to administration of trial drug or during the trial)
* Excessive physical activity within five days prior to administration of trial drug
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial centre
* marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
* Male subjects must agree to minimise the risk of female partners becoming pregnant from the dosing day until three months after the completion of the study. Acceptable methods of contraception for male volunteers include a vasectomy no less than three months prior to dosing, barrier contraception, or a medically accepted contraceptive method. For female partners of male volunteers, acceptable methods of contraception include intrauterine device, tubal ligation, hormonal contraceptive for at least two months, or diaphragm with spermicide
* Participation in more than one other radiolabelled investigational drug trial within one year prior to administration of the trial drug. The previous radiolabelled trial drug must have been received more than six months prior to administration of the trial drug for this study, and the total exposure from this study and the previous study will be within the recommended levels considered safe (e.g., less than 5000 mrem whole body annual exposure)
* Irregular defecation pattern (less than one bowel movement a day)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2009-06; Primary Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Individual concentration-time profiles of [14C]-radioactivity in whole blood, plasma, saliva, urine, and faeces | up to 28 days
Individual concentration-time profiles of BI 201335 ZW in plasma and urine | up to 28 days
Rate and extent of excretion mass balance based on the total radioactivity in urine and faeces | up to 28 days
Elucidation of metabolite structures and identification of major metabolites in urine, faeces, and plasma in comparison with various animal species | up to 28 days
Cblood cell/Cplasma ratio of [14C]-radioactivity | up to 28 days
Measurement of the plasma protein binding of total [14C]-radioactivity in human plasma samples ex vivo | up to day 28
Cmax,ss (maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | up to day 28
tmax,ss (time from last dosing to maximum concentration of the analyte in plasma at steady state) | up to day 28
Cmin,ss (minimum concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | up to day 28
AUCτ,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ) | up to day 28
λz,ss (terminal rate constant of the analyte in plasma at steady state) | up to day 28
t1/2,ss (terminal half-life of the analyte in plasma at steady state) | up to day 28
MRTpo,ss (mean residence time of the analyte in the body at steady state after oral administration) | up to day 28
CL/F,ss (apparent clearance of the analyte in the plasma at steady state following multiple oral dose administration) | up to day 28
Vz/F,ss (apparent volume of distribution of the analyte during the terminal phase λz at steady state following oral administration) | up to day 28
Ae,urine,0-tz,ss (amount of analyte that is eliminated in urine at steady state from the time point 0 to time point tz) | up to day 28
fe,urine,t1-t2,ss (fraction of the analyte in % of dose that is eliminated in urine at steady state from the time point 0 to time point tz) | up to day 28
Ae,feces,t1-t2,ss (fraction of the analyte that is eliminated in faeces at steady state from time point 0 to time point tz) | up to day 28
fe,feces,0-tz,ss (fraction of the analyte eliminated in faeces at steady state from time point 0 to time point tz) | up to day 28
CLR,t1-t2,ss (renal clearance of the analyte at steady state from the time point 0 to time point tz) | up to day 28

SECONDARY OUTCOMES:
Number of patients with abnormal findings in physical examination | Baseline and day 28
Number of patients with clinically significant changes in vital signs (blood pressure, pulse rate) | Baseline, day 1, 10, 16 and 28
Number of patients with clinically significant changes in 12-lead electrocardiogram (ECG) | Baseline, day 1, 10, 16 and 28
Number of patients with clinically significant changes in clinical laboratory tests (haematology, clinical chemistry, urinalysis) | Baseline, day 10 and 28
Number of patients with adverse events | up to 28 days
Assessment of tolerability on a 4-point scale by the investigator | Day 28